CLINICAL TRIAL: NCT05209386
Title: Flexible Representation of Speech in the Supratemporal Plane
Brief Title: Flexible Representation of Speech
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Carnegie Mellon University (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Taylor Abel, Assistant Professor of Neurological Surgery; Pediatric Neurosurgeon, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY21090011; 1R21DC019217-01A1 (NIH)
Record Dates: First submitted 2022-01-12; First posted 2022-01-26 (Actual); Results first posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Epilepsy
Keywords: sEEG; Speech representation; Supratemporal plane
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient Participants (Experimental): This single-group study will recruit patients through the PI's clinical practice who are undergoing invasive neurophysiological monitoring (sEEG) with clinically necessary placement of electrodes in the supratemporal plane.
  All participants will complete the same behavioral response paradigms.
  Interventions: Behavioral: Dimension-Based Statistical Learning

INTERVENTIONS:
Behavioral: Dimension-Based Statistical Learning — Each participant will complete self-paced blocks of stimuli that will first establish a baseline for neural activity and behavioral responses with clear speech, and will then record responses for experimentally manipulated blocks to introduce 1) speech-in-noise and 2) a Canonical-Reverse block to model an "accent." Auditory stimuli will be adjusted to a comfortable level for each participant as determined by a calibration process completed by the participant. Each block involves listening to sound via earphones and making a categorical decision between initial consonants (/b/ or /p/) by tapping a button to indicate the word heard by the participant.

SUMMARY:
The overarching goal of this exploratory research is to understand the dynamic and flexible nature of speech processing in the human supratemporal plane. The temporal lobe has long been established as a region of interest in the speech perception and processing literature because it contains the auditory cortex. More recently, research has localized the supratemporal plane as an area that exhibits response specificity to acoustic properties of complex auditory signals like speech. The supratemporal plane, comprised of Heschl's gyrus, the planum polare, and the planum temporale, is capable of the rapid spectrotemporal analysis required to map acoustic information to linguistic representation. Neural activity in this area, however, is rarely studied directly because it is difficult to access with non-invasive measures like scalp electroencephalography (EEG). Capitalizing on the unique opportunity to access these areas via routine clinical stereoelectroencephalography (sEEG) in a patient population, this study seeks to understand how cortical responses reflect the diagnosticity of two acoustic-phonetic dimensions of interest and how responses rapidly and flexibly adapt to changes in listening demands. Examining how neural response to voice onset time (VOT) and fundamental frequency (F0) modulates as a function of perceptual weight carried in signaling phoneme categories, and identifying how changes in listening context shift perceptual weight, will provide invaluable data that indicates how speech processing flexibly adapts to short-term acoustic patterns.

DETAILED DESCRIPTION:
The purpose of this study is to understand the dynamic, flexible nature of speech processing as a function of perceptual weight applied to acoustic-phonetic dimensions within varying listening contexts and demands.

The specific aims of this study are as follows:

1. To establish the neural response to two acoustic-phonetic dimensions as a function of the perceptual weight they carry when signaling phoneme identity.

   Aim 1 will specifically evaluate responses to voice onset time (VOT) and fundamental frequency (F0). Data collected will provide a baseline response for participants.
2. To identify how experimental manipulation of listening context impacts perceptual weighting strategies of VOT and F0.

Aim 2 will evaluate modulation of neural response to the introduction of noise and the introduction of an "accent."

A secondary aim of this study is to use "control" electrodes, which are those placed in clinically necessary regions of the brain but outside of the region of interest for this study (supratemporal plane), to determine if additional regions of the brain are implicated in adaptive plasticity of speech processing.

Speech is the primary means by which we convey our needs, wants, and thoughts to others and the ability to process speech is crucial to our everyday functioning, as well as our ability to establish and maintain relationships. Impairments in speech processing have an undeniable negative impact on individuals and society. While habilitative and rehabilitative strategies exist that can improve auditory processing and quality of life, understanding the exact neural mechanism underlying the human brain's ability to process speech would contribute to a more well-defined means by which to target deficits. This study seeks to understand the regions of the brain involved in speech processing, how those regions analyze specific acoustic-phonetic dimensions, and how the system adapts to successfully process speech in different listening contexts.

Modern electrophysiological techniques have revolutionized research into activity in the human brain, allowing investigators to identify specific regions or patterns of activity associated with various behaviors and sensory experiences. sEEG recordings, which involve intracerebral measurements of neural activity using depth electrodes, are capable of providing unique access to regions of the brain that are otherwise inaccessible with less invasive measurements. Capitalizing on PI Abel's work with pediatric patients undergoing sEEG recording for localization of seizure foci or language mapping, this study will allow researchers to directly study activity in regions that have already been implicated in the literature as crucial to spectrotemporal analysis of complex acoustic signals like speech. These regions within the supratemporal plane (STP) include Heschl's gyrus, the planum polare, and the planum temporale, all of which are uniquely targeted via sEEG.

Existing literature in speech processing has indicated that the mapping of physical input (acoustic signal) to linguistic representation (identification of phonemes or words) is not a static process, but rather highly dependent on listening context. The auditory processing system regularly adapts to changes in signal quality, adverse listening conditions, and short-term deviations from expected and learned regularities in native language input by applying varying importance, or perceptual weight, to specific acoustic-phonetic parameters. This indicates the existence of adaptive plasticity in speech processing, yet existing neurophysiological models do not account for this flexibility in cortical response. Data from pilot EEG and sEEG studies demonstrated that high gamma activity in the STP and behavioral responses were graded by the perceptual weight given to two acoustic-phonetic dimensions, voice onset time (VOT) and fundamental frequency (F0).

The proposed study will contribute to existing knowledge by helping to establish a more detailed model of on-line cortical response and adaptation to changing acoustic signals. It is unique in its accounting for the role that perceptual weight of acoustic-phonetic dimensions play in signaling phonemes and making category-based judgments.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 15-25 years old
* Undergoing sEEG placement in the supratemporal plane for clinically necessary localization of epileptic foci or language mapping
* Fluent English speakers
* Cognition and speech-language skills within normal limits (as determined by evaluation prior to surgery)
* Normal or correct-to-normal visual acuity
* Normal hearing acuity in each ear (as determined by audiometric assessment)
* No history of autism or ADHD

Exclusion Criteria:

* Individuals with intellectual disabilities
* Abnormal epileptiform activity in the supratemporal plane
* Lack of fluent English comprehension/production
* Severe language or auditory-specific cognitive dysfunction
* History of autism or ADHD

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taylor J Abel, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The individual deidentified participant data intended to be shared include the individual participant data that underlie the results to be reported in published articles after deidentification.
  Other documents that will be made available include the study protocol and statistical analysis plan.
  Data will be available as soon as possible following publication, but no later than one year upon completion. There is no end date.
  IPD will be made available for any purpose via open access.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available as soon as possible, but no later than one year upon completion of the study.
Access Criteria: Our data will be made publicly available online as soon as possible. Data will be easily and widely accessible.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from PI Abel's clinical population of patients undergoing invasive monitoring (sEEG) for drug-resistant epilepsy at Children's Hospital of Pittsburgh between May 2022-May 2025.
Pre-assignment Details: As there is only a single experimental group in this study, all enrolled patients were assigned to Arm 1 (Patient Participants).
Period: Overall Study
Arm/Group | Patient Participants
Started | 48
Completed | 16
Not Completed | 32
Not completed — Withdrawal by Subject | 8
Not completed — Period of sEEG implant insufficient to collect complete behavioral task | 24

BASELINE CHARACTERISTICS:
Arm/Group | Patient Participants
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.62 (3.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Phoneme Categorization [Mean (Standard Deviation); unit: percent of stimuli classified as /p/] — Behavioral responses to 2 alternative forced choice task asking participants to categorize stimuli as either /b/ or /p/ during the canonical block (i.e., stimuli containing typical combinations of VOT and F0). Reported here as mean percent of stimuli classified as /p/ during the canonical block.
  percent of stimuli classified as /p/ | 81.5 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: Supratemporal Neural Response to Change in Acoustic-Phonetic Dimensions
Description: Neural activity will be measured via simultaneous EEG-sEEG monitoring in the supratemporal plane as indicated by high-gamma band activity in the electrical signal. Neural activity will be measured as participants listen to acoustic stimuli with gradually manipulated acoustic dimensions, fundamental frequency (F0) and voice onset time (VOT). The data reported here is the number of temporal lobe channels demonstrating significant encoding of change in acoustic dimension (F0 as VOT is held constant).
Time Frame: During sEEG-EEG recording sessions, up to 3 hours total
Population: Neural data from 3 participants was contaminated by noise and was thus excluded from analysis.
Measure: Count of Units; unit: sEEG Channels
Units Other Than Participants: sEEG Channels
Groups:
- Patient Participants: This single-group study will recruit patients through the PI's clinical practice who are undergoing invasive neurophysiological monitoring (sEEG) with clinically necessary placement of electrodes in the supratemporal plane.
  All participants will complete the same behavioral response paradigms.
  Dimension-Based Statistical Learning: Each participant will complete self-paced blocks of stimuli that will first establish a baseline for neural activity and behavioral responses with clear speech, and will then record responses for experimentally manipulated blocks to introduce a Canonical-Reverse block to model an "accent." Auditory stimuli will be adjusted to a comfortable level for each participant as determined by a calibration process completed by the participant. Each block involves listening to sound via earphones and making a categorical decision between initial consonants (/b/ or /p/) by tapping a button to indicate the word heard by the participant.
Arm/Group | Patient Participants
Number analyzed (Participants) | 13
Number analyzed (sEEG Channels) | 618
sEEG Channels | 17
Statistical Analysis 1: Comparison: Patient Participants; Test type: Other; Permutation-based clustering analysis was used to identify channels that significantly encode change in acoustic dimensions. For each channel, a sliding-window encoding model was built comparing evoked responses (z-scored voltages) to Canonical Block stimuli across varying F0 with fixed VOT. This analysis identified the n = 17 channels and time windows where neural responses differed according to change in F0

2. Primary Outcome: Behavioral Impact of Change in Acoustic-Phonetic Dimensions
Description: Behavioral responses in the form of a category judgment will be obtained as participants listen to acoustic stimuli in with gradually varying fundamental frequency (F0) and voice onset time (VOT). Participants will provide a behavioral response by indicating the phoneme perceived at the beginning of stimulus words (/b/ or /p/). Specifically, the outcome is reported as percent of stimuli classified as /p/ over varying F0 with VOT held constant.
Time Frame: During sEEG-EEG recording sessions, up to 3 hours total
Population: 2 participants were excluded because they performed <50% on catch trials (0 and 40 ms VOTs); 1 participant was excluded because of a data quality issue
Measure: Mean (Standard Error); unit: percent of stimuli classified as /p/
Arm/Group | Patient Participants
Number analyzed (Participants) | 13
percent of stimuli classified as /p/ | 37.4 (6.4)
Statistical Analysis 1: Comparison: Patient Participants; Test type: Other; p < 0.0001, t-test, 2 sided; t(20.45) = -5.8

3. Primary Outcome: Supratemporal Neural Response to Change in Listening Context
Description: Neural activity was measured via sEEG monitoring as indicated by high-gamma band activity in the electrical signal. Neural activity will be measured as participants listen to acoustic stimuli in accented speech. The un-transformed voltage represents the difference in electric potential between a specific electrode contact and the reference electrode contact; since we use a common average reference, that means it's the difference between a specific electrode contact and the mean voltage across all electrodes. We then z-score to characterize shifts from baseline activity (where z = 0) at a specific electrode, which is believed to measure changes in voltage due largely to post-synaptic currents. This is a mathematical transformation rather than a published scale or standardized assessment. More extreme z-scores (+ or -) indicate a greater change from baseline local neural activity; in other words, stimuli evoked greater activity in this region.
Time Frame: During sEEG-EEG recording sessions, up to 3 hours total
Population: Neural data from 3 participants were contaminated by noise and therefore excluded from analysis. Channels included in this analysis were only those that demonstrated significant encoding of acoustic features (F0).
Measure: Mean (Standard Error); unit: Difference in z-scored voltage
Units Other Than Participants: sEEG Channels
Arm/Group | Patient Participants
Number analyzed (Participants) | 13
Number analyzed (sEEG Channels) | 17
Difference in z-scored voltage | 0.55 (0.12)
Statistical Analysis 1: Comparison: Patient Participants; Test type: Other; p < 0.0001, Mixed Models Analysis; For interaction term (effect of interest): t(1016) = -2.7; Time-averaged neural responses across respective windows of significance were averaged for all stimuli with ambiguous VOT (Canonical and Reverse blocks) to provide trial-averaged responses. A single linear mixed-effects model was built with fixed effects of F0, condition/listening context (block), and their interaction, as well as a random effect (intercept only) of patient+channel. The effect of interest was the interaction term, indicating that neural responses to F0 varied according to listening context (block)

4. Primary Outcome: Behavioral Impact of Change in Listening Context
Description: Behavioral responses in the form of a category judgment will be obtained as participants listen to acoustic stimuli in a varied listening context: accented speech. Participants will provide a behavioral response by indicating the phoneme perceived at the beginning of stimulus words (/b/ or /p/). Specifically, the outcome is reported as the mean % of stimuli classified as /p/ with varying VOT and F0 relationships.
Time Frame: During sEEG-EEG recording sessions, up to 3 hours total
Population: as for outcome 2
Measure: Mean (Standard Error); unit: percent of stimuli classified as /p/
Arm/Group | Patient Participants
Number analyzed (Participants) | 13
percent of stimuli classified as /p/
  Low F0/Ambiguous VOT | 54.9 (6.3)
  High F0/Ambiguous VOT | 30.3 (6.0)
Statistical Analysis 1: Comparison: Patient Participants; The null hypothesis is that there is no effect of change in listening context on behavioral responses of participants; Test type: Other; p < 0.0001, Mixed Models Analysis; t(48) = -4.50

5. Secondary Outcome: Neural Response of Non-Regions of Interest to Change in Acoustic-Dimension
Description: as for outcome 1
Time Frame: During sEEG-EEG recording sessions, up to 3 hours total
Population: Neural data from 3 participants was contaminated by noise and was thus excluded from analysis.
Measure: Count of Units; unit: sEEG Channels
Units Other Than Participants: sEEG Channels
Arm/Group | Patient Participants
Number analyzed (Participants) | 13
Number analyzed (sEEG Channels) | 2088
sEEG Channels | 4
Statistical Analysis 1: Comparison: Patient Participants; Test type: Other; Permutation-based clustering analysis was used to identify channels in non-regions of interest that significantly encode change in acoustic dimensions. For each channel, a sliding-window encoding model was built comparing evoked responses (z-scored voltages) to Canonical Block stimuli across varying F0 with fixed VOT. This analysis identified the n = 4 channels and time windows where neural responses differed according to change in F0

6. Secondary Outcome: Neural Response of Non-Regions of Interest to Change in Listening Context
Description: as for outcome 3
Time Frame: During sEEG-EEG recording sessions, up to 3 hours total
Population: Channels included in this secondary analysis (n = 4 from n = 3 patients) were only those that demonstrated significant encoding of acoustic features (F0).
Measure: Mean (Standard Error); unit: Difference in z-scored voltage
Units Other Than Participants: sEEG Channels
Groups:
- Patient Participants: This single-group study will recruit patients through the PI's clinical practice who are undergoing invasive neurophysiological monitoring (sEEG) with clinically necessary placement of electrodes in the supratemporal plane.
  All participants will complete the same behavioral response paradigms.
  Dimension-Based Statistical Learning: Each participant will complete self-paced blocks of stimuli that will first establish a baseline for neural activity and behavioral responses with clear speech, and will then record responses for experimentally manipulated blocks to introduce 1) speech-in-noise and 2) a Canonical-Reverse block to model an "accent." Auditory stimuli will be adjusted to a comfortable level for each participant as determined by a calibration process completed by the participant. Each block involves listening to sound via earphones and making a categorical decision between initial consonants (/b/ or /p/) by tapping a button to indicate the word heard by the participant.
Arm/Group | Patient Participants
Number analyzed (Participants) | 3
Number analyzed (sEEG Channels) | 4
Difference in z-scored voltage | -0.11 (0.064)
Statistical Analysis 1: Comparison: Patient Participants; Test type: Other; p = 0.480, Mixed Models Analysis; For interaction term (effect of interest): t(216) = -0.707; [other analysis details as in outcome 3, analysis 1]

ADVERSE EVENTS:
Time Frame: From enrollment until end of active participation in the behavioral task, on average 30-40 minutes.
Arm/Group | Patient Participants
All-Cause Mortality (participants affected / at risk) | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48
Other Adverse Events (participants affected / at risk) | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/86/NCT05209386/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-15): https://cdn.clinicaltrials.gov/large-docs/86/NCT05209386/SAP_001.pdf
  • Informed Consent Form (2022-07-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT05209386/ICF_002.pdf